CLINICAL TRIAL: NCT01322204
Title: Absorption and Metabolism of Oral Codeine in Mechanically Ventilated Neonates
Brief Title: Codeine in Mechanically Ventilated Neonates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jacob Aranda, Principal Investigator, State University of New York - Downstate Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10922
Record Dates: First submitted 2011-03-22; First posted 2011-03-24 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Mechanically Ventilated Neonates; Painful Procedures in Newborns
Keywords: codeine, neonates, pediatric pharmacology
MeSH Terms: interventions — Codeine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Neonates 0-30 days, no more than 2,000 grams, receiving mechanical ventilation.
  Interventions: Drug: Codeine

INTERVENTIONS:
Drug: Codeine — One single oral dose of 1 mg/kg of codeine

SUMMARY:
The purpose of this study is to determine the absorption and bioavailability of codeine in relation to postnatal (PNA) and postconceptional (PCA) age; determine the parent drug (codeine), its active metabolites, their formation rates and their ratios in relation with PCA and PNA; and identify relevant genetic polymorphisms of opioid metabolism in the study population and their potential relationship to the biodisposition and pharmacodynamic effects of codeine. The study population is intubated and mechanically ventilated infants equal to or greater than 26 weeks gestational age at birth and less than 4 weeks postnatal age.

DETAILED DESCRIPTION:
This proposal has its origins in a larger initiative to elucidate the pharmacological basis for the interindividual differences observed in opioid responsiveness. Gaps in our knowledge related to opioid disposition in newborns need to be addressed to complete the design of the required overarching initiative in which age could be treated as a continuous variable within a context of PK, PD and PG determinants.This proposal is designed to generate preliminary data that addresses two issues. First, can newborns absorb enterally administered codeine and is this ability determined by PCA or PNA age? The second relates to the ability of newborn infants to catalyze those reactions required to metabolically activate both codeine and morphine. The latter will also be evaluated within the context of PCA versus PNA age.

These data will not only fill an information gap that must be addressed before the larger initiative moves forward, but they also provide a platform for serious study of the ontogeny of certain pharmacokinetic processes that may prove critical to our understanding of newborn drug disposition. In this way, codeine can provide important insights concerning the ontogeny of drug disposition and permit the determination of the relative importance of PCA versus PNA ages to the functional expression of these processes.

ELIGIBILITY:
Inclusion Criteria:

* Neonates ≥ 26 weeks PCA receiving mechanical ventilation and painful procedure will be eligible for participation in the study
* Subject's parent/legal guardian must give written informed consent prior to study participation
* Subject is receiving opioid analgesia therapy based on caregiver determination. The ideal patient will not be receiving morphine.
* Must be able to receive an enteral dose of codeine.

Exclusion Criteria:

* Known hypersensitivity to morphine, fentanyl, or codeine
* Patients with ALT concentrations >2x upper limit of normal for age or clinical evidence of hepatic failure
* Patients with serum creatinine concentrations >2x upper limit of normal for age or clinical evidence of renal failure
* Patients who are NPO
* Babies born to maternal drug abuse.
* Total serum bilirubin level of > 10 mg/dl or 170 umol/L.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2008-08; Primary Completion 2013-03-06 (Actual); Study Completion 2013-03-06 (Actual)

PRIMARY OUTCOMES:
The rate and extent of absorption of oral codeine, the ratios of the observed concentration of each metabolite to the observed concentration of parent drug and the formation and clearances of the metabolites. | 2 hours

SECONDARY OUTCOMES:
Secondary outcomes include the additional PK parameters elimination half life, area under the curve and mean residence time. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jacob V Aranda, MD, PhD, Principal Investigator — State University of New York Downstate
Locations (1):
- State University of New York Downstate, Brooklyn, New York, United States